CLINICAL TRIAL: NCT03833648
Title: UControlPain App (This is the Official IRB Title)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18-1118
Record Dates: First submitted 2019-02-05; First posted 2019-02-07 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Opioid Use
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to one of two conditions: 1) usual care versus 2) provision of the provider-prescribed education/tool part of the consumer health informatics app (UControlPain) using a random electronic 1:1 allocation scheme.
Who Masked: Participant
Masking Description: Study participants will not know which version of the app they are instructed to install.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Usual Care (No Intervention): No intervention, patients will receive treatment as usual. Patients will download the UControl Pain app on their personal cell phones and will complete the four study surveys via the app or via REDCap.
- Arm 2 - UControl Pain App with Education (Experimental): Patients will install the UControl Pain app on their personal cell phones. The app will include educational information about pain management, e.g., using acetaminophen and NSAIDs for pain, as well as information on addiction and safe storage of medications. Subjects will also complete the four study surveys via the app or via REDCap.
  Interventions: Other: UControl Pain App with Education

INTERVENTIONS:
Other: UControl Pain App with Education — The intervention will include educational information on pain management, e.g., using acetaminophen and NSAIDs to manage pain, as well as information on addiction and safe storage of medications.
  Arms: Arm 2 - UControl Pain App with Education

SUMMARY:
It is estimated that 77% of all Americans own a smartphone and the use of health apps has doubled in the last two years. Consistent with this development, over half of US smartphone owners have downloaded a health-related mobile app. While patient engagement is an integral and well-established component of in-hospital Early Recovery After Surgery (ERAS) programs that drive improved perioperative outcomes, efforts to support such engagement are often limited to a patient's hospital stay. The objective of this aim is to empower patients to control their use of pain medications after surgery in a safe and effective fashion using a novel and innovative consumer health informatics app: UControlPain. This app will be leveraged to integrate three critical components of the study into one application: First, study recruitment and consent documentation. Second, application of the intervention engaging patients to take control of their pain management after discharge. Lastly, UControlPain will collect relevant patient outcomes including pain assessments, functional status, and quantification of opioid and non-opioid analgesic medication intake. Use of the app will reduce the amount of opioid medication required, while enhancing patient post-operative pain control by maximizing non-opioid therapy. Subjects will be able to employ flexible non-opioid therapy with acetaminophen and NSAIDs whenever possible and safe. The rationale is that testing of such a provider-prescribed consumer health informatics app (UControlPain) will lay the groundwork to scale this project towards more secure and efficient pain management practices after surgery on a systems level and beyond. Upon completion, the expectation is to have developed an effective consumer health informatics app to help patients better manage their post-surgical pain at home, reduce reliance on opioids, and improve opioid safety through enhanced storage and disposal behaviors.

DETAILED DESCRIPTION:
Prescription opioid overdose has emerged as a leading cause of death in the general population. Opioid-based therapy represents a corner-stone of post-operative pain management. With increasing emphasis on robust pain therapy, sales of opioid medications have increased. Parallel to this rise, opioid-associated deaths have also increased. Over-prescribed opioids after surgery can create a reservoir of opioids that become available for non-medical use. Effective strategies to maximize non-opioid pain therapy and to limit such a reservoir are lacking. Thus, there is an urgent need to individualize post-operative pain therapy and reduce reliance on opioids.

Preliminary data indicate that postsurgical patients are prescribed combination preparations (opioid+acetaminophen) in 96% of cases. Opioid+acetaminophen combination products have received scrutiny from the FDA for causing liver injury from unintentional overdose when combined with additional over-the-counter (OTC) acetaminophen. If postoperative patients are prescribed opioid-only products, they can safely use OTC acetaminophen in addition to NSAIDs, e.g. ibuprofen, in a highly effective fashion. Such an Alternatives to Opioids (ALTO)-based approach can reduce the need for opioids while ensuring pain control and limiting opioid-associated side effects. A barrier to utilizing an ALTO-based approach is lack of patient knowledge on appropriate use and timing of drugs such as acetaminophen, especially when used in combination with other analgesics. Internet-based applications have been successfully used for substance use disorder treatment adherence. Importantly, patient-based interventions to improve adherence are especially effective in the first six weeks, yielding up to five-fold improvement in compliance. While consumer health informatics applications have been successfully tested to improve adherence for anti-depressants and diabetic medications such an approach has not yet been evaluated for perioperative pain therapy. Data from an ongoing observational study assessing pain outcomes and patient-reported pain medication intake after hospital discharge support the assumption that effective combinations of non-opioid pain medications (ALTO) are underutilized.

The study is using an investigator engineered a functioning prototype of a consumer health informatics app: UControlPain. This study is a randomized controlled pilot trial of this consumer health informatics app, to test its effect on pain outcomes, analgesic medication requirements, and patient functional outcomes. For this study, the UControlPain will be introduced to hospitalized patients after surgery.

Patients will be approached regarding interest in the study prior to hospital discharge. A trained member of the research team will explain the study to prospective participants. If the patient is interested in participation the consent will be reviewed with the patient and the study team will answer any questions the patient may have. Then the study staff will assist the patient in downloading the UControlPain app. The study patient will be provided with a hard copy of the consent/HIPAA form.

Demographics and the best contact information will be collected from those enrolled patients who indicate they are interested in completing the surveys after their hospital discharge. Patients will be randomized to one of two conditions: 1) usual care versus 2) provision of the provider-prescribed education/tool part of the consumer health informatics app (UControlPain) using a random electronic 1:1 allocation scheme. If indicated and approved by the provider, opioid-only prescriptions will be written for opioid-based analgesia in both groups. Final dosing decisions and drug choices will remain at the discretion of the treating provider and nursing staff administering medications. While hospitalized patients will also be prompted to do a 6-minute walk test and measure the number of steps taken within 24 hours (if cleared by Physical Therapy to walk without assistance). These functional assessments will be performed daily while hospitalized and weekly for 4 weeks after discharge.

One week after hospital discharge interested patients with be contacted and asked to complete the first of four surveys. All communication will be available in English. Patients will be paid with a $5 gift card or money order equivalent to complete the study assessments within the app or with an online link.

UControlPain will provide general education on how to properly use ALTO, e.g., over-the-counter medications before using opioids in patients where providers have not identified contraindications to such medications (e.g. acetaminophen and non-steroidal anti-inflammatory drugs). Other educational information presented in this part of the app will include information on safe-storage, signs of overdose, and resources for patients who are concerned about becoming addicted. The survey part of the study consists of a brief questionnaire asking about pain management following hospital discharge that will be sent out weekly x 4 starting one week after hospital discharge.

ELIGIBILITY:
We will study up to 120 adult surgical patients, with the aim of having usable data from at least 90 patients.

Inclusion Criteria: 1) Patients ages 18-89 undergoing inpatient surgery at the University of Colorado Hospital are eligible. 2) Technical capacity and willingness to use and download the UControlPain app on their personal cell phone.

Exclusion Criteria: 1) Patients under the age of 18 years, 2) Patients returning to institutional settings (e.g. prison, jail, mental health facility), 3) Pregnant women, 4) Decisionally challenged patients, 5) Blind or illiterate patients, and 6) Medical contraindications to use of opioids, acetaminophen, or NSAIDs.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Mean Post-Discharge Opioid Intake at 4 weeks post-discharge (total) | Four weeks after hospital discharge, as reported on the surveys completed by the patient.
  Milligram morphine equivalent (MME)

SECONDARY OUTCOMES:
6-minute Walk Test - Week 1 | One week after hospital discharge
  Steps taken in a 6-minute walk test
6-minute Walk Test - Week 2 | Two weeks after hospital discharge
  Steps taken in a 6-minute walk test
6-minute Walk Test - Week 3 | Three weeks after hospital discharge
  Steps taken in a 6-minute walk test
6-minute Walk Test - Week 4 | Four weeks after hospital discharge
  Steps taken in a 6-minute walk test
In-Hospital Opioid Milligram Morphine Equivalent (MME) | 24 hours prior to hospital discharge
  Total MME of all in-hospital opioid medications prescribed in the 24 hours prior to hospital discharge as recorded in the electronic medical record (EMR) for each patient.
Mean Post-Discharge Opioid Dose | At the time of discharge
  Mean oral morphine equivalent (MME) post-discharge opioid dose
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Week 1 | One week after hospital discharge, as reported on the Week 1 survey completed one time by the patient.
  Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Score as reported on the Week 1 study survey. The Scale consists of 8 questions; each question in the Scale has five response options ranging in value from one to five, e.g., Not at all (1), A little bit (2), Somewhat (3), Quite a bit (4), Very much (5). To find the total raw score sum the values of the response to each question. The lowest possible raw score is 8; the highest possible raw score is 40, with a lower score indicating a better outcome/less pain interference. Raw scores are then translated into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Week 2 | Two weeks after hospital discharge, as reported on the Week 2 survey completed one time by the patient.
  Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Score as reported on the Week 2 study survey. The Scale consists of 8 questions; each question in the Scale has five response options ranging in value from one to five, e.g., Not at all (1), A little bit (2), Somewhat (3), Quite a bit (4), Very much (5). To find the total raw score sum the values of the response to each question. The lowest possible raw score is 8; the highest possible raw score is 40, with a lower score indicating a better outcome/less pain interference. Raw scores are then translated into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Week 3 | Three weeks after hospital discharge, as reported on the Week 3 survey completed one time by the patient.
  Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Score as reported on the Week 3 study survey. The Scale consists of 8 questions; each question in the Scale has five response options ranging in value from one to five, e.g., Not at all (1), A little bit (2), Somewhat (3), Quite a bit (4), Very much (5). To find the total raw score sum the values of the response to each question. The lowest possible raw score is 8; the highest possible raw score is 40, with a lower score indicating a better outcome/less pain interference. Raw scores are then translated into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Week 4 | Four weeks after hospital discharge, as reported on the Week 4 survey completed one time by the patient.
  Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Score as reported on the Week 4 study survey. The Scale consists of 8 questions; each question in the Scale has five response options ranging in value from one to five, e.g., Not at all (1), A little bit (2), Somewhat (3), Quite a bit (4), Very much (5). To find the total raw score sum the values of the response to each question. The lowest possible raw score is 8; the highest possible raw score is 40, with a lower score indicating a better outcome/less pain interference. Raw scores are then translated into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Week 1 | One week after hospital discharge, as reported on the Week 1 survey completed one time by the patient.
  Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Score as reported on the Week 1 study survey. The Scale consists of 3 questions; each question in the Scale has five response options ranging in value from one to five, e.g., No pain (1), Mild (2), Moderate (3), Severe (4), Very Severe (5). To find the total raw score sum the values of the response to each question. The lowest possible raw score is 3; the highest possible raw score is 15, with a lower score indicating a better outcome/less pain intensity. Raw scores are then translated into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Week 2 | Two weeks after hospital discharge, as reported on the Week 2 survey completed one time by the patient.
  Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Score as reported on the Week 2 study survey. The Scale consists of 3 questions; each question in the Scale has five response options ranging in value from one to five, e.g., No pain (1), Mild (2), Moderate (3), Severe (4), Very Severe (5). To find the total raw score sum the values of the response to each question. The lowest possible raw score is 3; the highest possible raw score is 15, with a lower score indicating a better outcome/less pain intensity. Raw scores are then translated into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Week 3 | Three weeks after hospital discharge, as reported on the Week 3 survey completed one time by the patient.
  Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Score as reported on the Week 3 study survey. The Scale consists of 3 questions; each question in the Scale has five response options ranging in value from one to five, e.g., No pain (1), Mild (2), Moderate (3), Severe (4), Very Severe (5). To find the total raw score sum the values of the response to each question. The lowest possible raw score is 3; the highest possible raw score is 15, with a lower score indicating a better outcome/less pain intensity. Raw scores are then translated into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Week 4 | Four weeks after hospital discharge, as reported on the Week 4 survey completed one time by the patient.
  Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Score as reported on the Week 4 study survey. The Scale consists of 3 questions; each question in the Scale has five response options ranging in value from one to five, e.g., No pain (1), Mild (2), Moderate (3), Severe (4), Very Severe (5). To find the total raw score sum the values of the response to each question. The lowest possible raw score is 3; the highest possible raw score is 15, with a lower score indicating a better outcome/less pain intensity. Raw scores are then translated into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Non-opioid pain medications taken | One week after hospital discharge, as reported on the Week 1 survey completed one time by the patient.
  Mean doses in milligrams
Non-opioid pain medications taken | Two weeks after hospital discharge, as reported on the Week 2 survey completed by the patient.
  Mean doses in milligrams
Non-opioid pain medications taken | Three weeks after hospital discharge, as reported on the Week 3 survey completed by the patient.
  Mean doses in milligrams
Non-opioid pain medications taken | Four weeks after hospital discharge, as reported on the Week 4 survey completed by the patient.
  Mean doses in milligrams

OTHER OUTCOMES:
Opioid storage and disposal | Hospital discharge until 4 weeks after discharge
  Locked vs. un-locked location

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Bartels, MD, PhD, Principal Investigator — CU Anschutz Medical Campus
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. Aggregate data may be shared with other researchers as required by some journals or as requested by qualified investigators as determined by the study PI. However, the names and any other personal health information that identifies research subjects will always be kept confidential and will not be shared.

REFERENCES:
- [Background] Milani RV, Franklin NC. The Role of Technology in Healthy Living Medicine. Prog Cardiovasc Dis. 2017 Mar-Apr;59(5):487-491. doi: 10.1016/j.pcad.2017.02.001. Epub 2017 Feb 11. PMID 28189614
- [Background] Krebs P, Duncan DT. Health App Use Among US Mobile Phone Owners: A National Survey. JMIR Mhealth Uhealth. 2015 Nov 4;3(4):e101. doi: 10.2196/mhealth.4924. PMID 26537656
- [Background] Liu VX, Rosas E, Hwang J, Cain E, Foss-Durant A, Clopp M, Huang M, Lee DC, Mustille A, Kipnis P, Parodi S. Enhanced Recovery After Surgery Program Implementation in 2 Surgical Populations in an Integrated Health Care Delivery System. JAMA Surg. 2017 Jul 19;152(7):e171032. doi: 10.1001/jamasurg.2017.1032. Epub 2017 Jul 19. PMID 28492816
- [Background] Centers for Disease Control and Prevention. Prescription Drug Overdose: Understanding the Epidemic. http://www.cdc.gov/drugoverdose/data/index.html Accessed last on 09/28/2017.
- [Background] Centers for Disease Control and Prevention. Leading Causes of Death. http://www.cdc.gov/injury/wisqars/leading_causes_death.html Accessed last on 09/27/2017.
- [Background] Acute Pain Management: Operative or Medical Procedures and Trauma. Agency for Healthcare Research and Quality (AHCPR). 1992; http://archive.ahrq.gov/clinic/medtep/acute.htm. Accessed 12/11/2014.
- [Background] Centers for Disease Control and Prevention (CDC). Vital signs: overdoses of prescription opioid pain relievers---United States, 1999--2008. MMWR Morb Mortal Wkly Rep. 2011 Nov 4;60(43):1487-92. PMID 22048730
- [Background] Volkow ND, Frieden TR, Hyde PS, Cha SS. Medication-assisted therapies--tackling the opioid-overdose epidemic. N Engl J Med. 2014 May 29;370(22):2063-6. doi: 10.1056/NEJMp1402780. Epub 2014 Apr 23. No abstract available. PMID 24758595
- [Background] Olsen Y, Daumit GL, Ford DE. Opioid prescriptions by U.S. primary care physicians from 1992 to 2001. J Pain. 2006 Apr;7(4):225-35. doi: 10.1016/j.jpain.2005.11.006. PMID 16618466
- [Background] Calcaterra S, Glanz J, Binswanger IA. National trends in pharmaceutical opioid related overdose deaths compared to other substance related overdose deaths: 1999-2009. Drug Alcohol Depend. 2013 Aug 1;131(3):263-70. doi: 10.1016/j.drugalcdep.2012.11.018. Epub 2013 Jan 5. PMID 23294765
- [Background] Binswanger IA, Blatchford PJ, Mueller SR, Stern MF. Mortality after prison release: opioid overdose and other causes of death, risk factors, and time trends from 1999 to 2009. Ann Intern Med. 2013 Nov 5;159(9):592-600. doi: 10.7326/0003-4819-159-9-201311050-00005. PMID 24189594
- [Background] Dart RC, Surratt HL, Cicero TJ, Parrino MW, Severtson SG, Bucher-Bartelson B, Green JL. Trends in opioid analgesic abuse and mortality in the United States. N Engl J Med. 2015 Jan 15;372(3):241-8. doi: 10.1056/NEJMsa1406143. PMID 25587948
- [Background] Bartels K, Fernandez-Bustamante A, McWilliams SK, Hopfer CJ, Mikulich-Gilbertson SK. Long-term opioid use after inpatient surgery - A retrospective cohort study. Drug Alcohol Depend. 2018 Jun 1;187:61-65. doi: 10.1016/j.drugalcdep.2018.02.013. Epub 2018 Mar 27. PMID 29627407
- [Background] Rodgers J, Cunningham K, Fitzgerald K, Finnerty E. Opioid consumption following outpatient upper extremity surgery. J Hand Surg Am. 2012 Apr;37(4):645-50. doi: 10.1016/j.jhsa.2012.01.035. Epub 2012 Mar 10. PMID 22410178
- [Background] Harris K, Curtis J, Larsen B, Calder S, Duffy K, Bowen G, Hadley M, Tristani-Firouzi P. Opioid pain medication use after dermatologic surgery: a prospective observational study of 212 dermatologic surgery patients. JAMA Dermatol. 2013 Mar;149(3):317-21. doi: 10.1001/jamadermatol.2013.1871. PMID 23682368
- [Background] Food and Drug Adminstration. Department of Health and Human Services. Prescription Products Containing Acetaminophen; Actions To Reduce Liver Injury From Unitentional Overdose. Federal Register. 2011;76(10):2691-2697.
- [Background] Derry CJ, Derry S, Moore RA. Single dose oral ibuprofen plus paracetamol (acetaminophen) for acute postoperative pain. Cochrane Database Syst Rev. 2013 Jun 24;2013(6):CD010210. doi: 10.1002/14651858.CD010210.pub2. PMID 23794268
- [Background] Valentine AR, Carvalho B, Lazo TA, Riley ET. Scheduled acetaminophen with as-needed opioids compared to as-needed acetaminophen plus opioids for post-cesarean pain management. Int J Obstet Anesth. 2015 Aug;24(3):210-6. doi: 10.1016/j.ijoa.2015.03.006. Epub 2015 Mar 23. PMID 25936786
- [Background] Barozzi N, Tett SE. Perceived barriers to paracetamol (acetaminophen) prescribing, especially following rofecoxib withdrawal from the market. Clin Rheumatol. 2009 May;28(5):509-19. doi: 10.1007/s10067-008-1077-8. Epub 2009 Jan 9. PMID 19132456
- [Background] Campbell AN, Nunes EV, Matthews AG, Stitzer M, Miele GM, Polsky D, Turrigiano E, Walters S, McClure EA, Kyle TL, Wahle A, Van Veldhuisen P, Goldman B, Babcock D, Stabile PQ, Winhusen T, Ghitza UE. Internet-delivered treatment for substance abuse: a multisite randomized controlled trial. Am J Psychiatry. 2014 Jun;171(6):683-90. doi: 10.1176/appi.ajp.2014.13081055. PMID 24700332
- [Background] Sirey JA, Banerjee S, Marino P, Bruce ML, Halkett A, Turnwald M, Chiang C, Liles B, Artis A, Blow F, Kales HC. Adherence to Depression Treatment in Primary Care: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Nov 1;74(11):1129-1135. doi: 10.1001/jamapsychiatry.2017.3047. PMID 28973066